CLINICAL TRIAL: NCT05374772
Title: A Retrospective, Real World Study to Analyze Disease Outcomes in Patients With Mild to Moderate Coronavirus Disease 2019 (COVID-19)
Brief Title: A Retrospective Study in Patients With Mild to Moderate COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Pudong Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: JT001-011-COVID-19
Record Dates: First submitted 2022-05-13; First posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: COVID-19
Keywords: Mild to Moderate COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with COVID-19: Mild to moderate COVID-19 patient with at least one risk factor for serve COVID-19 illness or death.

SUMMARY:
The purpose of this retrospective study is to analyze real-world disease progression in mild-moderate COVID-19 patients with at least one risk factor for serve COVID-19 illness or death.

DETAILED DESCRIPTION:
This study is a retrospective, real world study, without any intervention in clinical diagnosis and treatment, and only real world data are collected for analysis.

The investigator will review symptoms, risk factors, and other non-invasive inclusion and exclusion criteria.

The study will collect and analyze available symptoms, risk factors and SARS-COV-2 Ct value up to 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have a positive SARS-CoV-2 test result.
* Participants who have one or more mild or moderate COVID-19 symptoms.
* Participants who have one or more of the following requirements: ≤7 days from the first positive test for SARS-COV-2 virus infection to Day 1; ≤5 days from the first onset of COVID-19 symptoms to Day 1.
* Participants who satisfy one or more than one of the following high risks for progression to severe COVID-19, including death.

Exclusion Criteria:

* Participants who are diagnosed with severe/critical COVID-19 before Day 1.
* Participants who have SpO2≤93% on room air at sea level or PaO2/FiO2≤ 300, or respiratory rate ≥30 per minute before Day 1.
* Participants who have received mechanical ventilation before Day 1.
* Participants who have received or plan to receive a SARS-CoV-2 monoclonal antibody treatment or prevention, or antiviral treatment (including the investigational treatment) before and during hospitalization.
* Participants who have received convalescent COVID-19 plasma treatment before and during hospitalization.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Mild to Moderate COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-05-13 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of the participants who have progression of COVID-19 | Day 1 to 28 days
  Percentage of participants who experience these events: Progress to severe and/or critical COVID-19; Death from any cause
Percentage of participants who experience these events | Day 1 to 28 days
  Percentage of participants who experience these events: Progress to severe and/or critical COVID-19; Death from any cause

SECONDARY OUTCOMES:
Time to sustained clinical recovery | Up to 28 days
  Time to sustained clinical recovery
Time to sustained disappearance of clinical symptoms | Up to 28 days
  Time to sustained disappearance of clinical symptoms
Time to initial negative conversion of SARS-COV-2 | Up to 28 days
  Time to initial negative conversion of SARS-COV-2
Time to sustained negative conversion of SARS-CoV-2 | Up to 28 days
  Time to sustained negative conversion of SARS-CoV-2
Percentage of participants who turned negative for SARS-CoV-2 | Day 3, 5, 7, 10, 14
  Percentage of participants who turned negative for SARS-COV-2 at Day 3, 5, 7, 10, 14
The change of SARS-COV-2 Ct value | Day 3, 5, 7, 10, 14
  The change of SARS-COV-2 Ct value The change of SARS-COV-2 Ct value at Day 3, 5, 7, 10, 14
Safety assessment Results: such as AEs and SAEs through Day 28 | Up to 28 days
  Safety assessment Results: such as AEs and SAEs through Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Minghua Yu, Principal Investigator — Shanghai Pudong Hospital
Locations (1):
- Shanghai Pudong Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No